CLINICAL TRIAL: NCT06223035
Title: Identification of Exercise-induced Myokines Regulating the Muscle-adipose Signaling Axis
Brief Title: Myokine Identification Following Acute Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LOL-1044
Record Dates: First submitted 2023-11-30; First posted 2024-01-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Secretome characterization and signaling to the adipose tissue (Experimental): To identify possible exercise stimulated secreted proteins which signal to the adipose tissue, subcutaneous adipose and blood will be collected both before and at multiple timepoints following a VO2max test. Adipose will be collected from the abdominal subcutaneous region and blood will be collected from the arm. Blood will be analyzed for change in protein abundance and adipose will be analyzed for change in gene expression.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will take part in a VO2max test. This will include a graded exercise test (GXT) on a motorized treadmill while wearing a one-way, non-rebreathing valve and nose clip that allows for the evaluation of all expired air. Specifically, we will incorporate the Ellestad Protocol. The Ellestad Protocol is divided into 8 phases which gradually increases in speed and incline throughout the test. The VO2max test will continue until the participant reaches volitional fatigue defined by reaching a rate of perceived exertion (RPE) greater than 19 (using the Borg RPE Scale), OR a respiratory exchange ratio (RER) reaching above 1.1, OR a participant choosing to cease exercise for any reason.

SUMMARY:
Exercise stimulates a cascade of responses within the human body. For example, exercise results in the release of proteins into the circulation which communicate with cells and organs throughout the body. In fact, recent human research identified more than 600 proteins are released into the blood circulation following short-term exercise, many of which are predicted to come from the skeletal muscle and target the fat tissue. However, identification of these muscle-secreted proteins and their target tissue (i.e. fat tissue) remains extremely challenging. This challenge is because tissue needs to be collected from multiple sites (skeletal muscle and fat) and at multiple timepoints (before and after exercise). This study seeks to address these challenges through the collection of fat and blood both before and after short-term exercise followed by protein detection (of the blood) and gene expression (of the fat tissue).

DETAILED DESCRIPTION:
Acute exercise stimulates a cascade of responses within the human body. Not only do tissues work in an autonomous manner, but they also secrete factors mediating interorgan communication. Recent human research identified >600 proteins secreted into the circulation following an acute bout of exercise, many of which are predicted to derive from the skeletal muscle and target the adipose tissue. Indeed, human studies have validated the effect exercise-induced myokines have upon adipose physiology, most notably IL-6. While insightful, identification of myokines and their tissue of target (i.e. adipose tissue) remains extremely challenging in humans. This is largely due to the need for tissue collection from multiple sites (skeletal muscle and adipose tissue) and at multiple timepoints (before and after exercise). To address these challenges, This study will implement an acute bout of exercise in a human cohort, followed by tissue collection and in-depth secretome and tissue protein analysis. This study will accomplish these goals through tissue and blood collection at multiple timepoints before and after exercise followed by in-depth proteome and transcriptome analysis.

For the first in-person visit, participants will arrive to The Rockefeller University Hospital between 8:00am to 10:00am in a non-fasted state. All participants will be asked to keep track of their food consumption both the night prior to and the day of the visit. Participants will be asked to consume their breakfast 2-hours prior to arrival, and will be asked to eat their habitual breakfast. Participants will be asked to refrain from intense physical activity 48 hours prior to the testing day, any caffeinated beverages the day of arrival, and any alcoholic beverages for 24-hours prior to arrival.

Height, weight, resting heart rate, blood pressure, and body composition, will be measured. Blood will be collected from the upper arm for blood chemistry analyses including HbA1c (%), Cholesterol (mg/dl), LDL-cholesterol (mg/dl), HDL-cholesterol (mg/dl), Triglyceride (mg/dl), Complete blood count (CBC), and High sensitivity C-reactive protein (hsCRP). An additional 20mL of blood will be drawn from the arm for protein identification through the use of proteomics. Subcutaneous adipose from the lower abdomen will be collected following blood collection.

Following a minimum of one week from fat sample collection, participants will take part in a maximal aerobic consumption (VO2max) test between 8:00am-10:00am. Participants will arrive in a non-fasted state, but all participants will be asked to keep track of their food consumption the night prior to, and the morning of, the VO2max test. When possible, the investigators will recommend the participants to consume the identical dinner/breakfast to that consumed prior to the first in-person visit. Participants will be asked to consume their breakfast 2-hours prior to arrival. Additionally, participants will be asked to refrain from intense physical activity 48 hours prior to the testing day, any caffeinated beverages the day of arrival, and any alcoholic beverages for 24-hours prior to arrival.

For VO2max testing, participants will take part in a general warm up consisting of walking on a motorized treadmill for 5 minutes followed by performing a graded exercise test (GXT) on a motorized treadmill while wearing a one-way, non-rebreathing Hans Rudolph 7450 series V2 mask that allows for the evaluation of all expired air which is calibrated prior to each test. Volume of ventilated expired air as well as oxygen and carbon dioxide concentrations of expired air will be determined using a commercial metabolic cart (Parvo Medics' TrueOne® 2400, Parvo, UT). Specifically, the investigators will incorporate the Ellestad Protocol to determine the participants VO2max. The Ellestad Protocol is divided into 8 phases which gradually increases in speed and incline throughout the test. To confirm that the VO2max test is eliciting a metabolic response, lactate measurements through the use of a finger prick will be taken both before and immediately following the exercise test. Additionally, participants will wear a light-weight heart rate monitoring device (Polar) strapped around the upper torso during testing to track heart rate throughout exercise.

The VO2max test will continue until the participant reaches volitional fatigue defined by reaching a rate of perceived exertion (RPE) greater than 19 (using the Borg RPE Scale), OR a respiratory exchange ratio (RER) reaching above 1.1, OR a participant choosing to cease exercise for any reason.

Blood will be collected from the arm immediately following exercise, 1-hour following the exercise, and 3-hours following exercise. Adipose will be collected Immediately following the final blood draw, participants will be prepped for adipose tissue collection (from the abdominal subcutaneous adipose). This will occur 3-hours following exercise.

ELIGIBILITY:
Inclusion Criteria:

* passing the PARQ questionnaire (i.e. answering "NO" to all questions)
* being between the ages of 18-45
* being moderately active (defined as participating in 30 minutes of recreational activity at least once per week for the past 3 months but no more than 3 times per week)
* non-smoking
* free of metabolic or cardiovascular diseases

Exclusion Criteria:

* unhealed fractures
* thrombophlebitis (blood clots)
* recent surgery of the upper or lower extremities (any surgeries in past 6 months at the ankle or foot, or in the past year at the knee, hip, shoulder or elbow)
* recent uncontrolled bruising
* recent muscle, bone or joint damage which interferes with regular physical activity
* taking part in vigorous physical activity more than 3 times per week
* any prior sensations of chest pain during exercise.
* individuals who are pregnant as determined by an on-site pregnancy test
* individuals who are currently taking exogenous hormones
* individuals who chronically consume NSAIDS or other anti-inflammatory medication (every day for the previous 3 months)
* failing the PARQ questionnaire as indicated by answering "YES" to any of the questions
* Having a BMI >32
* Any medical condition that in the opinion of the investigator will confound interpretation of data for analysis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Identification and quantification of exercise-induced proteins released into the blood through the use of proteomic analysis. | Before exercise, immediately following exercise, 1-hour following exercise, 3-hours following exercise
  The change in protein abundance within the circulation will be identified by using proteomic-based detection methods. Proteins detected from the control timepoint (before exercise), will be compared to the three timepoints following exercise.

SECONDARY OUTCOMES:
Characterize changes in gene expression of the subcutaneous adipose tissue following exercise through the use of bulk RNA-sequencing. | 1 week pre-intervention, 1-hour following, 3-hours following
  Bulk RNA-sequencing of subcutaneous adipose tissue will be analyzed both before and following acute exercise. The investigators will seek to identify those genes which show differential gene expression between the pre and post exercise timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Olsen, PhD, Principal Investigator — The Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker JM, Garcet S, Aleman JO, Mason CE, Danko D, Butler D, Zuffa S, Swann JR, Krueger J, Breslow JL, Holt PR. Obesity and ethnicity alter gene expression in skin. Sci Rep. 2020 Aug 21;10(1):14079. doi: 10.1038/s41598-020-70244-2. PMID 32826922